CLINICAL TRIAL: NCT00541918
Title: COGNITIVE - Comparison of Cognitive Function After Sevoflurane or Propofol Anesthesia for Open-heart Operations
Brief Title: COGNITIVE - Cognitive Function After Sevoflurane or Propofol Anesthesia for Open-heart Operations
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: study suspended due to staff indisposition
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Maciej M. Kowalik, Dr., Medical University of Gdansk
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: AMG-NKBEN/560/2006
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Other Functional Disturbances Following Cardiac Surgery; Memory Disorders
Keywords: sevoflurane,; propofol,; heart surgery,; cardiopulmonary bypass,; memory disorders,
MeSH Terms: conditions — Memory Disorders | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): propofol
  Interventions: Drug: Diprivan (propofol, Astra Zeneca)
- 2 (Experimental): sevoflurane
  Interventions: Drug: Sevorane (sevoflurane, Abbott)

INTERVENTIONS:
Drug: Diprivan (propofol, Astra Zeneca) — Total intravenous anesthesia with propofol
  Other Names: propofol
  Arms: 1
Drug: Sevorane (sevoflurane, Abbott) — inhaled anesthesia with sevoflurane
  Other Names: sevoflurane
  Arms: 2

SUMMARY:
The aim of the study is to prove whether general anesthesia with inhaled sevoflurane reduces the frequency of neurological and cognitive impairment after open-heart operations with use of cardiopulmonary by-pass (CPB) in comparison with intravenous anesthesia with propofol.

DETAILED DESCRIPTION:
Patients assigned to the "sevoflurane" group will be anesthetized with inhaled sevoflurane (induction and conduction of general anesthesia) and empirically administered fentanyl und pancuronium. During the CPB, sevoflurane will be delivered via the oxygenator of the CPB-machine.

Patients assigned to the "propofol" group will be anesthetized with continuous propofol infusion and empirically administered fentanyl and pancuronium.

The level of anesthesia will be monitored with BIS (bi-spectral index) - desirable level of 40 - 60.

Following preoperative data will be recorded: age, years of school education, NYHA-class, LVEF by TTE, comorbidities, glucosylated hemoglobin in patients with diabetes, non-invasive arterial blood pressure the day before the operation, smoked cigarettes, alcohol abuse.

Recorded data from operation: type of surgery, CBP duration, aortic clamp duration, duration of arterial hypotension (MAP < 60 mmHg) on CPB or SAP < 90 after CPB, the lowest perfusion gradient (MAP-CVP), the lowest pO2 in arterial blood and lowest blood oxygen saturation, lowest and average brain blood saturation (measured by INVOS), steroid dosis, aprotinin dosis, mannitol dosis on CPB, epiaortic echocardiography for aortic clamping, TEE before weaning from CPB with evaluation of deaeration of the left ventricle, highest serum glucose level, highest oesophageal temperature.

Data collected after operation: time to tracheal extubation, doses of catecholamines, consciousness disorders, CRP, S-100b protein, glucose level, core temperature, ICU stay, stay at the surgery department, hospital stay.

The patients will undergo a psychological examination four times: before the operation, before discharge from hospital (usually 4-6 days after the operation), 3 and 12 months after the operation. The psychological test for evaluating the cognitive modalities will include:

1. verbal learning - the Rey's AVLT test
2. direct verbal memory - number repeating attempt from the WAIS-R/PL test
3. direct nonverbal memory - Memory Test of Geometric Figures by Benton
4. operating memory test - TMT test
5. the cognitive interference test - a modified Stroop test
6. verbal fluence - according to the Boston Test of Aphasia
7. concentration and work effectiveness - by the Number Symbol test by Wechsler.
8. mood - Beck's depression scale
9. NEECHAM Delirium Scale - during the first 24-36 hours after surgery
10. the Gough's Adjective Test will be performed with in-house relatives of the patient for evaluation the eventual emotional and eventual personality changes

Neurological examination will be performed before and 6 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* adults
* valve-repair open-heart surgery without coronary artery bypass grafting

Exclusion Criteria:

* active infective endocarditis
* previous cardiac surgery
* emergency operations
* chronic renal failure (serum creatinine > 2,0 mg/dL)
* left ventricle ejection fraction < 30%
* myocardial infarction within last 30 days

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
results of psychological examination | 6 days, 3 and 12 months after surgery

SECONDARY OUTCOMES:
S-100B protein level in serum. NEECHAM delirium scale, stroke or other severe neurological impairment | S-100B - 18 hours after surgery; Consciousness and/or neurological impairment - within 6 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Romuald Lango, M.D., Ph.D., Study Director — Medical University of Gdańsk, Department of Cardiac Anesthesiology
Locations (2):
- Poland (2):
  - Department of Cardiac Anesthesiology, Medical University of Gdańsk, Gdansk
  - Medical Universty of Gdańsk, Department of Cardiac and Vascular Surgery, Gdansk

REFERENCES:
- See also: Home page of the Department of Cardiac Anesthesiology, MUG. — http://www.amg.gda.pl/uczelnia/informator/jednostka.php?id=327